CLINICAL TRIAL: NCT02524782
Title: A Phase 1, Combined Single- and Multiple-ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics (PK), and Pharmacodynamics (PD) of MEDI4166 in Subjects With Type 2 Diabetes Mellitus (T2D)
Brief Title: A Phase 1, Single- and Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of MEDI4166 in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D6240C00001
Record Dates: First submitted 2015-08-13; First posted 2015-08-17 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2018-03

CONDITIONS: Type 2 Diabetes
Keywords: MEDI-4166, diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MEDI-4166 (Experimental): MEDI-4166 administered subcutaneously
  Interventions: Biological: MEDI-4166
- Placebo (Placebo Comparator): Placebo administered subcutaneously
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: MEDI-4166 — MEDI-4166 administered subcutaneously
  Arms: MEDI-4166
Biological: Placebo — Placebo administered subcutaneously
  Arms: Placebo

SUMMARY:
A Phase 1, combined Single Ascending Dose (SAD) and Multiple-ascending Dose (MAD) study to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of MEDI4166 in Subjects with Type 2 Diabetes Mellitus (T2D).

DETAILED DESCRIPTION:
This study is a first time in human (FTIH), Phase 1, randomized, double-blind study to evaluate the safety, tolerability, PK, and PD of MEDI4166 administered as both single and multiple ascending doses to subjects with T2D.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes, ages 18-65
* Must provide written informed consent
* BMI>=25 and =<42
* Venous access suitable for multiple cannulations
* Vital signs within normal specified ranges
* Females must be non-lactating and non-childbearing potential
* Males must practice 2 effective contraceptive measures if sexually active

Exclusion Criteria:

* Any concurrent condition that in the opinion of the investigator would interfere with the evaluation of the investigational product
* History or presence of gastrointestinal, renal, or hepatic disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs
* History of cancer, with the exception of basal cell carcinoma or carcinoma of the cervix
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks prior to dosing
* Positive Hepatitis B, Hepatitis C or HIV test or use of antiretroviral medications at screening
* Current or previous use of systemic corticosteroids within the past 28 days prior to screening
* Use of any medicinal products or herbal preparations licensed for weight loss is prohibited.
* Positive drug screen
* Type 1 diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2015-10-07 (Actual); Primary Completion 2017-04-14 (Actual); Study Completion 2017-04-14 (Actual)

PRIMARY OUTCOMES:
Part A: Number of subjects with adverse events as a measure of safety and tolerability of MEDI4166 | 43 days post dosing
  Treatment emergent adverse events (TEAEs) and serious adverse events (TESAEs)
Part A: Number of subjects with adverse events as a measure of safety and tolerability of MEDI4166 | 43 days post dosing
  12 lead electrocardiogram including RR, PR, QRS, QT and QTc intervals
Part A: Number of subjects with adverse events as a measure of safety and tolerability of MEDI4166 | 43 days post dosing
  Vital signs (systolic and diastolic blood pressure, pulse rate, temperature, and respiratory rate)
Part A: Number of subjects with adverse events as a measure of safety and tolerability of MEDI4166 | 43 days post dosing
  Clinical laboratory assessments (serum chemistry, hematology, urinalysis)
Part A: Number of subjects with adverse events as a measure of safety and tolerability of MEDI4166 | 43 days post dosing
  Physical examination
Part B: Change in glucose AUC measured up to 240 minutes after mixed meal tolerance test (MMTT) from baseline to Day 36 | 36 days post dosing
  Part B: Change in glucose AUC measured up to 240 minutes after mixed meal tolerance test (MMTT) from baseline to Day 36
Part B: Change in LDL-C from baseline to Day 36 | 36 days post dosing
  Part B: Change in LDL-C from baseline to Day 36

SECONDARY OUTCOMES:
Part A: Pharmacokinetics of MEDI4166, maximum plasma concentration (Cmax) | 43 days post dosing
  Part A: Pharmacokinetics of MEDI4166, maximum plasma concentration (Cmax)
Part A: Pharmacokinetics of MEDI4166, area under the curve concentration (AUC) | 43 days post dosing
  Part A: Pharmacokinetics of MEDI4166, area under the curve concentration (AUC)
Part A: Change from baseline in LDL-C | 43 days post dosing
  Part A: Change from baseline in LDL-C
Part A: Proportion of subjects with Anti-drug Antibodies (ADA) to MEDI4166 | 43 days post dosing
  Part A: Proportion of subjects with ADA to MEDI4166
Part B: Number of subjects with adverse events as a measure of safety and tolerability of MEDI4166 | 71 days post dosing
  Treatment emergent adverse events (TEAEs) and serious adverse events (TESAEs)
Part B: Number of subjects with adverse events as a measure of safety and tolerability of MEDI4166 | 71 days post dosing
  12 lead electrocardiogram including RR, PR, QRS, QT and QTc intervals
Part B: Number of subjects with adverse events as a measure of safety and tolerability of MEDI4166 | 71 days post dosing
  Vital signs (systolic and diastolic blood pressure, pulse rate, temperature, and respiratory rate)
Part B: Number of subjects with adverse events as a measure of safety and tolerability of MEDI4166 | 71 days post dosing
  Clinical laboratory assessments (serum chemistry, hematology, urinalysis)
Part B: Number of subjects with adverse events as a measure of safety and tolerability of MEDI4166 | 71 days post dosing
  Physical examination
Part B: Pharmacokinetics of MEDI4166, maximum plasma concentration (Cmax) | 71 days post dosing
  Part B: Pharmacokinetics of MEDI4166, maximum plasma concentration (Cmax)
Part B: Pharmacokinetics of MEDI4166, area under the curve concentration (AUC) | 71 days post dosing
  Part B: Pharmacokinetics of MEDI4166, area under the curve concentration (AUC)
Part B: Change from baseline in fructosamine levels | 36 days post dosing
  Part B: Change from baseline in fructosamine levels
Part B: Proportion of subjects with ADA to MEDI4166 | 71 days post dosing
  Part B: Proportion of subjects with ADA to MEDI4166
Part A: Pharmacokinetics of MEDI4166, time to maximum observed plasma drug concentration (Tmax) | 43 days post dosing
  Part A: Pharmacokinetics of MEDI4166, time to maximum observed plasma drug concentration (Tmax)
Part A: Change from baseline in glucose AUC up to 240 minutes | 43 days post dosing
  Part A: Change from baseline in glucose AUC up to 240 minutes
Part B: Pharmacokinetics of MEDI4166, time to maximum observed plasma drug concentration (Tmax) | 71 days post dosing
  Part B: Pharmacokinetics of MEDI4166, time to maximum observed plasma drug concentration (Tmax)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Research Site, Anniston, Alabama
  - Research Site, Chula Vista, California
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, South Miami, Florida
  - Research Site, Durham, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Knoxville, Tennessee
  - Research Site, San Antonio, Texas

REFERENCES:
- [Derived] Jain M, Carlson G, Cook W, Morrow L, Petrone M, White NE, Wang T, Naylor J, Ambery P, Lee C, Hirshberg B. Randomised, phase 1, dose-finding study of MEDI4166, a PCSK9 antibody and GLP-1 analogue fusion molecule, in overweight or obese patients with type 2 diabetes mellitus. Diabetologia. 2019 Mar;62(3):373-386. doi: 10.1007/s00125-018-4789-6. Epub 2018 Dec 28. PMID 30593607